CLINICAL TRIAL: NCT02477995
Title: Study of Adsorption Tetanus-diphtheria-acellular Pertussis (DTaP) Vaccine in Healthy Infants 3 to 5 Months of Age: A Randomized, Blinded, Single-center, Positive Controlled Clinical Trial
Brief Title: Study of Adsorption Tetanus-diphtheria-acellular Pertussis (DTaP) Vaccine in Healthy 3 to 5 Months Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1110103
Record Dates: First submitted 2015-06-09; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2011-07

CONDITIONS: Pertussis
Keywords: Immunogenicity; Safety; DTaP Vaccine
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DTaP Vaccine A (Experimental): Adsorption tetanus-diphtheria-acellular pertussis (DTaP) Vaccine A(Bejing minhai Biological Co., LTD) of 0.5ml in 600 infants aged 3-5months on day 0, 28, 56.
  Interventions: Biological: DTaP Vaccine A
- DTaP Vaccine B (Active Comparator): Adsorption tetanus-diphtheria-acellular pertussis (DTaP) Vaccine B (Changchun changsheng Biological Co., LTD ) of 0.5ml in 600 infants aged 3-5months on day 0, 28, 56.
  Interventions: Biological: DTaP Vaccine B

INTERVENTIONS:
Biological: DTaP Vaccine A — Adsorption tetanus-diphtheria-acellular pertussis (DTaP) Vaccine A(Bejing minhai Biological Co., LTD) of 0.5ml, three doses, 28 days interval
  Arms: DTaP Vaccine A
Biological: DTaP Vaccine B — Adsorption tetanus-diphtheria-acellular pertussis (DTaP) Vaccine B(Changchun changsheng Biological Co., LTD ) of 0.5ml in 600 infants aged 3-5months on day 0, 28, 56.
  Arms: DTaP Vaccine B

SUMMARY:
Pertussis, diphtheria and tetanus are seriously infectious diseases in children. Since using of the adsorption diphtheria-tetanus-whole-cell pertussis (DTwP), it greatly reduced incidence of the three kinds of diseases. But the thallus of pertussis in the vaccine may cause more side reactions after vaccination. Since 2000, the basic immunization DTwP vaccine has been replaced by adsorption tetanus-diphtheria-acellular pertussis vaccine in American. In 1995, DTaP was successfully developed in China, and have been used in EPI at present. Because of effective immunity and little side reaction, DTaP has been widely recognized and accepted by the parents.

DETAILED DESCRIPTION:
Pertussis, diphtheria and tetanus are seriously infectious diseases for children. The world health organization (WHO) included the adsorption diphtheria-tetanus-whole-cell pertussis (DTwP) into the expanded program on immunization (EPI), as a basic immunization. Since using the DTwP, it greatly reduced incidence of the three kinds of diseases. Thousands of children have been saved since its application. Although the DTwP was productively in against pertussis, diphtheria and tetanus, thallus of pertussis in the vaccine could cause more side reactions after vaccination. Many individuals did not want to be vaccinated. However, there was two large epidemics of pertussis during the period of 1977-1979 and 1981-1983. Since 2000, the basic immunization DTwP vaccine has been replaced by adsorption tetanus-diphtheria-acellular pertussis vaccine (DTaP) vaccine in American. In 1995, DTaP was successful developed in the investigators' country, and is used in EPI at present. Because of effective immunity and causing little side reaction, DTaP has been widely recognized and accepted by the parents. This clinical trial is planning to evaluate the immunogenicity and safety of DTaP in 3-5 months infants .

ELIGIBILITY:
Inclusion criteria:

* Healthy infants aged 3-5months old as established by medical history and clinical examination
* The subjects' guardians are able to understand and sign the informed consent
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature ≤37.0°C on axillary setting

Exclusion criteria:

* Subjects who was premature birth
* Subjects who has a medical history of diphtheria, pertussis or tetanus.
* Had been vaccined for DTwP or DTaP
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Severe malnutrition or dysgenopathy
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Thyroid disease
* Coagulation disorder diagnosed by a doctor(such as the lack of clotting factors, clotting hemorrhagic disease, platelet abnormalities) or significant bruising
* No spleen, functional asplenia, and any situation caused by no spleen or splenectomy
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids
* Any prior administration of blood products in last 3 month
* Any prior administration of other research medicines in last 1 month
* Any prior administration of attenuated live vaccine in last 15 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Had fever before vaccination, Subjects with temperature >37.0°C on axillary setting
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Exclusion criteria for the second and third dose:

If subjects who have one condition of 1 to 4 as followed, prohibiting to continue the vaccination, and they will be continue observed in the opinion of the investigator. If Subjects who had one condition of 5 to 6 as followed, must be determined whether to continue by the investigator. If Subjects who had one condition of 7 to 8 as followed, they can had a delayed vaccination during time frame of the program. All participants with adverse events as followed, must be settled in follow-up to the end of events.

* Any serious adverse events caused by vaccination.
* Hypersensitivity after vaccination.
* Anaphylaxis after vaccination
* Any confirmed or suspected autoimmune diseases or immune deficiency disorders, including human immunodeficiency virus (HIV) infection
* Have acute or new chronic disease during vaccination
* Other reactions that in the opinion of the investigator ( include: severely serious symptom of pain, swelling, Limitation of motion, continuous high fever, headache and other Systemic or local reactions )
* Have acute disease during vaccination (Acute disease refers to with or without fever of moderate or severe disease)
* Subjects with temperature >37.0°C on axillary settin.

Ages: 3 Months to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity after vaccination | Day 28 post-dose 3
  The seroconversion rate of anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibody on day 28 post-dose 3.
  seroconversion is defined as post-third dose anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibody concentrations ≥ protective antibody concentration, if pre-vaccination concentration is < protective antibody concentration or ≥ 4 x protective antibody concentration if pre- vaccination concentrations ≥ protective antibody concentration.
Proportion of subjects reporting solicited injection-site reactions, solicited systemic reactions. | Day 7 post-each dose
  Proportion of subjects reporting solicited injection-site reactions, solicited systemic reactions on day 7 post-each dose.

SECONDARY OUTCOMES:
The seropositivity rates of anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibodies in serum on day 28 post-dose3. | Day 28 post-dose 3
  The seropositive rates of anti-pertussis tox oid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibodies in serum on day 28 post-dose3. Seropositivity is defined as post-third dose anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibody concentrations ≥ protective antibody concentration.
Proportion of subjects reporting unsolicited injection-site and systemic reactions. | Day 28 post-each dose
Proportion of subjects with serious adverse events(SAE) occurring throughout the trial. | Day 0 up to 90 post-vaccination
Geometric mean concentration(GMC)of anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibodies in serum on day 28 post-dose3. | Day 28 post-dose 3
Geometric mean fold increase（GMFI）of anti-pertussis toxoid , anti- filamentous hemagglutinin, anti-diphtheria toxoid and anti-tetanic antibodies in serum on day 28 post-dose3. | Day 28 post-dose 3

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Bachelor, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China